CLINICAL TRIAL: NCT01634087
Title: A Double-Blind, Placebo-Controlled Study Exploring the Safety, Tolerability, and Efficacy of a 28-Day Course of Escalating Doses of Oral Itacitinib in Subjects With Stable, Chronic Plaque Psoriasis
Brief Title: A Study of Escalating Doses of Itacitinib Administered Orally in Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 39110-250
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — itacitinib; INCB039110

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 100 mg QD Itacitinib (Experimental)
  Interventions: Drug: Itacitinib
- 100 mg QD Placebo (Experimental)
  Interventions: Drug: Placebo
- 200 mg QD Itacitinib (Experimental)
  Interventions: Drug: Itacitinib
- 200 mg QD Placebo (Experimental)
  Interventions: Drug: Placebo
- 200 mg BID Itacitinib (Experimental)
  Interventions: Drug: Itacitinib
- 200 mg BID Placebo (Experimental)
  Interventions: Drug: Placebo
- 600 mg once a day Itacitinib (Experimental)
  Interventions: Drug: Itacitinib
- 600 mg once a day Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Itacitinib — Itacitinib administered orally
  Other Names: INCB039110
  Arms: 100 mg QD Itacitinib; 200 mg BID Itacitinib; 200 mg QD Itacitinib; 600 mg once a day Itacitinib
Drug: Placebo — Placebo administered orally
  Arms: 100 mg QD Placebo; 200 mg BID Placebo; 200 mg QD Placebo; 600 mg once a day Placebo

SUMMARY:
This is a study of itacitinib in patients with chronic plaque psoriasis. This study will evaluate safety and efficacy parameters of itacitinib.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic plaque psoriasis aged 18 to 75 who have had insufficient response to topical agents, and who meet the psoriasis assessment expectations as defined in the study protocol

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Men and women who cannot comply with requirements to avoid fathering a child or becoming pregnant, respectively
* Subjects treated with leflunomide or other biological therapies to treat psoriasis and all JAK-STAT inhibitors within 12 weeks prior to first dose of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of itacitinib as measured by changes in frequency and severity of adverse events, ECGs, physical examination, vital signs, and clinical laboratory evaluations. | Approximately two months.
The mean percent change from baseline in static Physician's Global Assessment (sPGA) on the day 28 visit. | Approximately 28 days.

SECONDARY OUTCOMES:
Percentage of subjects achieving static Physician's Global Assessment (sPGA) of 1 or 2 at each scheduled visit. | Day 1, Day 8, Day 15, Day 28 and Day 56 (approximately two months).
Preliminary Pharmacokinetic (PK) collections. | Following 15 days of therapy.
  Plasma concentrations of itacitinib will be used to estimate peak plasma concentration (Cmax) and area under the plasma concentration-time curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Victor Sandor, MD, Study Director — Incyte Corporation
Locations (9):
- United States (5):
  - Hot Springs, Arkansas
  - Los Angeles, California
  - Clinton, Minnesota
  - Fridley, Minnesota
  - Rochester, New York
- Canada (4):
  - Moncton, New Brunswick
  - Windsor, Ontario
  - Montreal, Quebec
  - Québec